CLINICAL TRIAL: NCT01374503
Title: A Phase I, Single-centre, Randomised, Single-blinded, Placebo-controlled Single Ascending Dose Study, Followed by an Open-label Extension, Evaluating the Safety, Pharmacokinetics, Pharmacodynamics and Efficacy of ALX-0651, Administered Intravenously to Healthy Male Volunteers
Brief Title: First in Man Study of ALX-0651, a Nanobody Inhibiting CXCR4
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Proof of principle established with completed SAD part
Sponsor: Ablynx, a Sanofi company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALX-0651-1.1/11
Record Dates: First submitted 2011-06-14; First posted 2011-06-16 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALX-0651 (Experimental)
  Interventions: Biological: ALX-0651
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ALX-0651 — single or multiple (once daily for maximum 3 consecutive days) i.v. administration, 0.003-12 mg/kg
  Arms: ALX-0651
Biological: Placebo — single or multiple i.v. administration
  Arms: Placebo

SUMMARY:
The purpose of this first-in-man Phase I study is to determine whether the CXCR4-inhibitor ALX-0651 is safe and effective after single or multiple intravenous administrations to healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers, aged >= 18 and <= 55 at screening.
* Willing to consent to using an effective contraceptive method for at least 3 months after test substance administration.
* Non-smokers, or ex-smokers abstinent from tobacco for at least 1 year.
* Body mass index (BMI): 19 - 29 kg/m2 (extremes included).
* Haematology and chemistry parameters within normal range or showing no clinically relevant deviations, as judged by the Medical Investigator. For haematology, haemoglobin and white blood cell (WBC) count must be within normal limits. For chemistry, calcium, alkaline phosphatase (ALP), (alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma-glutamyl transferase (GGT) and lactate dehydrogenase (LDH) must be within normal limits.
* Normal electrocardiogram, showing no clinically relevant deviations, as judged by the Investigator. QTc <= 450 ms.
* No history or presence of diseases of the kidneys, heart, lungs, liver, gastrointestinal tract or endocrine organs, or other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* No history of clinically relevant allergies.
* Obtained, signed and dated informed consent.
* Ability and willingness to comply with protocol requirements.

Exclusion Criteria:

* Intake of any prescribed systemic or topical medication within 14 days prior to dosing.
* Intake of vitamin A derivates or retinoids within 30 days prior to the start of drug administration.
* History of thrombosis.
* Chronic infection or acute significant infection or fever within the last 5 weeks prior to the start of test substance administration.
* Subjects with any abnormality of the spleen (confirmed by echography) or history of splenic disease, or subjects that underwent splenectomy in the past.
* Blood donation (>500 ml) or a comparable blood loss within three months prior to the start of drug administration.
* Subjects who, in the investigator's opinion, may not be capable of following the study schedule for any reason, with special emphasis on eligibility for the aphaeresis procedure.
* Participation in an investigational drug study within 60 days prior to drug administration, or within less than 6 times the terminal elimination half-life of the test substance used in the respective trial (whichever is longer).
* Malignancy, or prior malignancy, with a disease-free interval of < 5 years after diagnosis and intervention, except curative treatment for non-melanoma skin cancer or resected carcinoma in situ.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2011-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events | until 1 month after study drug administration

SECONDARY OUTCOMES:
maximum plasma concentration (Cmax) of ALX-0651 | from predose until 48 hours after study drug administration
  Plasma concentration of ALX-0651 will be determined at different timepoints between predose and 48 hours after the last study drug administration. The maximum plasma concentration (Cmax) of ALX-0651 will be derived from the resulting plasma concentration versus time plots.
CD34 positive cell count in blood | from predose until 14 days after study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Josefin-Beate Holz, MD, Study Director — Ablynx NV
Locations (1):
- Groningen, Netherlands